CLINICAL TRIAL: NCT01978769
Title: The Effect of Physical Effort in the Decision Making Process of Preadolescents With ADHD
Status: Completed | Type: Observational
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: effortdiscounting.ctil
Record Dates: First submitted 2013-07-11; First posted 2013-11-08 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2013-07

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Preadolescents with ADHD: preadolescents with prior diagnosis of ADHD and without any other psychiatric or neurological diagnosis.
- Preadolescents with out any diagnosis: Preadolescents with out any diagnosis

SUMMARY:
In the current study we will examine a specific aspect of these processes that has yet to be studied. We will test the effect that a physically effortful assignment has on the choices that a preadolescent makes using a forced choice paradigm in which the participant will be asked to choose between and carry out either a high cost-high reward option (HR) or a low cost-low reward (LR) option. The HR option will demand a significant amount of physical effort and will be paired up with a large reward as opposed to the LR option which will be less demanding physically and paired up with a small reward. The assignment will be carried out using a hand held dynamometer which measures the power produced by the participants' upper extremity.

We propose that a child with attention deficit hyperactivity disorder (ADHD) will choose a task that involves less effort despite the small reward tied to it compared to a control child who will choose the more demanding task and the larger reward.

DETAILED DESCRIPTION:
In the current study we will examine a specific aspect of these processes that has yet to be studied. We will test the effect that a physically effortful assignment has on the choices that a preadolescent makes using a forced choice paradigm in which the participant will be asked to choose between and carry out either a high cost-high reward option (HR) or a low cost-low reward (LR) option. The HR option will demand a significant amount of physical effort and will be paired up with a large reward as opposed to the LR option which will be less demanding physically and paired up with a small reward. The assignment will be carried out using a hand held dynamometer which measures the power produced by the participants' upper extremity.

We propose that a child with ADHD will choose a task that involves less effort despite the small reward tied to it compared to a control child who will choose the more demanding task and the larger reward.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of ADHD

Exclusion Criteria:

* any other neurological or psychiatric diagnosis

Ages: 11 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: residents of jerusalem
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2014-11; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
The number of "low effort" choices of the ADHD participants compared to the number of "low effort" choices of the control participants | immediately after testing

CONTACTS AND LOCATIONS:
Overall Officials: yehuda polak, Dr., Principal Investigator — Hebrew University of Jerusalem
Locations (1):
- Shaarei Zedek Medical Center, Jerusalem, Israel, Israel